CLINICAL TRIAL: NCT07291934
Title: Effect of Pilates and Resistance Training on Pain, Disability, and Sleep Quality in Patients With Chronic Low Back Pain and Sleep Disturbances
Brief Title: Pilates and Resistance Training for Pain, Disability, and Sleep in Chronic Low Back Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Mosab ALdabbas, ASSISTANT PROFESSOR AT AL AZHAR UNIVERSITY, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: ALAZHAR UNIVERSITY in Gaza
Record Dates: First submitted 2025-12-05; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Chronic Low Back Pain
Keywords: sleep; chronic low back pain; disability; Pilate; Resistance traning
MeSH Terms: interventions — Resistance Training; Exercise Movement Techniques

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Combined Intervention Group (Pilates + Resistance Training): (Experimental): Participants in this group will receive both Pilates and resistance training exercises. The program will be supervised 2 times per week for 8 weeks.This arm is designed to evaluate the synergistic effect of the combined interventions on pain, disability, and sleep quality.
  Interventions: Other: Combined Intervention (Pilates + Resistance Training)
- Pilates Group (Experimental): Participants will perform Pilates exercises only under supervision 2 times per week for 8 weeks, with optional home practice. This arm will assess the effectiveness of Pilates alone on the study outcomes.
  Interventions: Other: Pilates
- Control Group (Usual Care): (Other): Participants in the control group will continue their routine care without structured or supervised exercise. This group will serve as a baseline comparison to determine the effects of the interventions beyond standard care.
  Interventions: Other: Control (Usual Care)

INTERVENTIONS:
Other: Combined Intervention (Pilates + Resistance Training) — Participants will receive both Pilates and resistance training exercises, supervised 2 times per week for 8 weeks. This intervention aims to evaluate the combined effect on improving pain, disability, and sleep quality.
  Arms: Combined Intervention Group (Pilates + Resistance Training):
Other: Pilates — Participants will perform Pilates exercises only, supervised 2 times per week for 8 weeks. This intervention will assess the effectiveness of Pilates alone on the study outcomes.
  Arms: Pilates Group
Other: Control (Usual Care) — Participants will continue their routine care without structured exercise. This intervention serves as a baseline comparison to determine the effects of the exercise programs beyond standard care.
  Arms: Control Group (Usual Care):

SUMMARY:
This study will investigate the effect of Pilates and resistance training on pain, disability, and sleep quality in patients with chronic low back pain and sleep disturbances. Participants will be randomly assigned into three groups:

Combined intervention group: Pilates plus resistance training

Single intervention group: Pilates alone

Control group: Advices only

All interventions will be delivered 3 times per week for 8 weeks, with outcome measures assessed at baseline, post-intervention (8 weeks), and follow-up (16 weeks). It is expected that the combined intervention group will show the greatest improvements in pain, disability, and sleep quality, while the single intervention group will demonstrate moderate benefits compared with usual care.

DETAILED DESCRIPTION:
This study will investigate the effects of Pilates and resistance training on pain, disability, and sleep quality in patients with chronic low back pain and sleep disturbances in the Gaza Strip. The study will use a 3-arm randomized controlled trial design, with participants randomly assigned to one of three groups:

Combined Intervention Group: Pilates plus resistance training

Single Intervention Group: Pilates or resistance training alone

Control Group: Usual care

The intervention groups will participate in 2 supervised sessions per week for 8 weeks. The control group will continue their usual care without structured or supervisedexercise.

Outcome measures will be assessed at baseline, post-intervention (8 weeks), and follow-up (16 weeks). The outcomes include pain intensity and disability, while sleep quality.

The study aims to determine whether the combined exercise intervention produces greater improvements than a single exercise intervention or usual care, providing evidence for the most effective rehabilitation strategy for patients with chronic low back pain and sleep disturbances.

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed with chronic low back pain (CLBP), defined as pain localized between the lower rib margin and gluteal folds, lasting ≥12 weeks.
* Sleep Quality: Poor sleep quality, defined as PSQI global score >5.

Exclusion Criteria:

* Specific LBP causes: Low back pain due to fractures, tumors, infections, inflammatory disorders, or systemic disease.
* Recent spinal surgery: History of lumbar spine surgery within the past 12 months.
* Severe comorbidities: Serious cardiovascular, respiratory, neurological, or musculoskeletal disorders that contraindicate exercise.
* Pregnancy or planned pregnancy during the study period.
* Current participation in structured exercise programs targeting the back (Pilates, resistance training, or core stabilization) within the last 3 months.
* Use of sleep medications or interventions that cannot be maintained stable during the study period.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 110 (Estimated)
Dates: Start 2026-01-25 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity: | Assessment Time Points: Baseline (pre-intervention) Post-intervention (8 weeks) Follow-up (16 weeks)
  Measured using the Visual Analog Scale (VAS), a 10-cm line where 0 indicates "no pain" and 10 indicates "worst imaginable pain." It captures the patient's perceived pain severity.
Disability | Assessment Time Points: Baseline (pre-intervention) Post-intervention (8 weeks) Follow-up (16 weeks)
  Oswestry Disability Index (ODI)
  The Oswestry Disability Index (ODI) is a widely used, validated questionnaire that assesses functional disability in individuals with low back pain. It measures the impact of back pain on a person's ability to perform activities of daily living (ADL) and overall functional limitations.
  Structure:
  The ODI contains 10 sections, each focusing on a different aspect of daily function:
  Pain intensity
  Personal care (washing, dressing)
  Lifting
  Walking
  Sitting
  Standing
  Sleeping
  Social life
  Traveling
  Employment/homemaking
  Each section has 6 statements scored from 0 to 5, with higher scores indicating greater disability.
Sleep_ Pittsburgh Sleep Quality Index (PSQI) | Assessment Time Points: Baseline (pre-intervention) Post-intervention (8 weeks) Follow-up (16 weeks)
  The Pittsburgh Sleep Quality Index (PSQI) is a validated, self-reported questionnaire used to assess sleep quality and disturbances over the past month. It is widely used in clinical and research settings, including studies on chronic pain and musculoskeletal disorders.
  Structure:
  The PSQI consists of 19 individual items combined into 7 components:
  Subjective sleep quality - the individual's perception of their sleep
  Sleep latency - time taken to fall asleep
  Sleep duration - total hours of sleep per night
  Habitual sleep efficiency - percentage of time in bed actually spent sleeping
  Sleep disturbances - factors causing sleep interruptions (e.g., waking up, pain, environmental disturbances)
  Use of sleep medication - frequency of taking sleep aids
  Daytime dysfunction - difficulty staying awake or maintaining function during the day
  Scoring:
  Each component is scored from 0 (no difficulty) to 3 (severe difficulty).
  The component scores are summed to generate a global PSQI score

IPD SHARING:
Plan to Share IPD: No